CLINICAL TRIAL: NCT03044197
Title: Assessing the Detection of Clinically Significant Prostate Cancer Using Magnetic Resonance Imaging-Guided Transperineal Targeted Biopsy Compared to Standard Transrectal Biopsy Outcomes Study: The ASTROS Trial
Brief Title: Detection of Clinically Significant Prostate Cancer Using Transperineal Targeted Biopsy Compared to Standard Transrectal Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0013
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer; Magnetic Resonance Imaging; Target Lesion; Fusion Biopsy; Clinically Significant Prostate Cancer; Transperineal
Keywords: prostate cancer; magnetic resonance imaging; transperineal biopsy; target lesion; fusion biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Erythema Multiforme

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to arm A or arm B following a 1:1 simple randomization procedure according to a computer-generated randomization list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MRI/ultrasound transperineal prostate biopsy (Experimental): In arm A, all patients with positive mpMRI evidence of lesions suspicious for PCa, i.e. PI RADS ≥ 3 will be submitted to transperineal mpMRI-targeted prostate biopsy (arm A MRI+). The gland and the regions of interest will be contoured, and the prostate contour will be fused in real time with the TRUS image. Biopsies will be performed via a transperineal approach in the operating room. The patient will be placed in dorsal lithotomy position. mpMRI-targeted biopsies will be performed on regions of interest, and three to six cores will be obtained for biopsy from each lesion and is standard of care according to START criteria for targeted biopsy. In cases of negative mpMRI results i.e. PI RADS<3, arm A patients will undergo TRUS-guided transrectal 12-core prostate biopsy (arm A MRI-) as described in arm B.
  Interventions: Device: MRI/ultrasound transperineal prostate biopsy
- transrectal ultrasound-guided prostate biopsy (Active Comparator): TRUS-guided transrectal prostate biopsy will be performed using a disposable 18-gauge biopsy gun with a specimen size of 18-22 mm (Bard Medical, Covington, GA, USA). The 12 cores will be obtained from 12 separate anatomical regions of the prostate which is standard practice in performing TRUS-guided transrectal prostate biopsy: left medial apex, left lateral apex, left medial midgland, left lateral midgland, left medial base, left lateral base, right medial apex, right lateral apex, right medial midgland, right lateral midgland, right medial base and right lateral base.
  Interventions: Device: transrectal ultrasound-guided prostate biopsy

INTERVENTIONS:
Device: MRI/ultrasound transperineal prostate biopsy — 3-6 targeted biopsy cores from each prostate region of interest
  Arms: MRI/ultrasound transperineal prostate biopsy
Device: transrectal ultrasound-guided prostate biopsy — 12 systematic biopsy cores
  Arms: transrectal ultrasound-guided prostate biopsy

SUMMARY:
Prostate biopsies are currently the gold standard for the diagnosis of prostate cancer. Many biopsies, however, are unnecessary or cannot detect significant prostate cancer (PCa). With multi-parametric magnetic resonance imaging (mpMRI) we now potentially have a way of increasing the detection of detecting clinically significant prostate cancer (csPCa) while decreasing the detection of non-significant PCa.

DETAILED DESCRIPTION:
In men with previously negative prostate biopsy and persistent elevated prostate-specific antigen (PSA) value, it is unclear which biopsy strategy offers the highest detection rate for significant prostate cancer. The hypothesis of this study is that targeted MRI/ultrasound fusion-guided biopsy improves the detection rates of clinically significant prostate cancers (csPCa) compared with systematic transrectal ultrasound-guided prostate biopsy.

Patients who fulfill all eligibility criteria and have provided written consent will be randomized to undergo MRI followed by biopsies (arm A) or TRUS transrectal biopsy (arm-B). Patients will be randomly assigned to arm A or arm B following a 1:1 simple randomization procedure according to a computer-generated randomization list. The primary end point will be the comparison of detection rates csPCa between arm A and arm B. csPCa will be defined according to the Standards of Reporting for MRI-targeted Biopsy Studies (START) criteria for targeted biopsy Gleason Score ≥ 7 or maximum CCL ≥ 5 mm and the updated Epstein criteria for SB (Gleason score ≥ 7, PSA density ≥ 0.15, Gleason score ≥ 2 positive cores, and bilateral cancer). The secondary end points will be (1) Comparison of the overall detection rate of PCa and csPCa between arm A mpMRI+ and arm B and (2) Comparison of complication rates between arm A mpMRI+ and arm B.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18-75 years old
2. PSA >1 ng/ml but <15 ng/ml
3. Negative DRE
4. Signed informed consent

Exclusion Criteria:

1. Previous prostate biopsy or prostate surgery
2. Previous prostate mpMRI
3. Contraindication to mpMRI: patients with pacemakers, defibrillators or other implanted electronic devices
4. Patients in the Texas Department of Criminal Justice (prisoners)
5. Patients with acute urinary symptoms including urinary retention and urinary tract infection

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Williams, MD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch at Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kosarek CD, Mahmoud AM, Eyzaguirre EJ, Shan Y, Walser EM, Horn GL, Williams SB. Initial series of magnetic resonance imaging (MRI)-fusion targeted prostate biopsy using the first transperineal targeted platform available in the USA. BJU Int. 2018 Nov;122(5):909-912. doi: 10.1111/bju.14206. Epub 2018 Apr 14. PMID 29569311

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI/Ultrasound Transperineal Prostate Biopsy | Transrectal Ultrasound-guided Prostate Biopsy
Started | 12 | 12
Completed | 9 | 11
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: 3 subjects in Arm A and 1 subject in Arm B withdrew from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI/Ultrasound Transperineal Prostate Biopsy | Transrectal Ultrasound-guided Prostate Biopsy | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Full Range); unit: years] — Population: 3 subjects in Arm A and 1 subject in Arm B withdrew from the study.
  years | 64 [56 to 71] | 60 [54 to 68] | 62 [54 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Prostate Cancer
Description: Number of subjects with positive clinically significant prostate cancer results
Time Frame: Within 2-4 wks after biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | MRI/Ultrasound Transperineal Prostate Biopsy | Transrectal Ultrasound-guided Prostate Biopsy
Number analyzed (Participants) | 9 | 11
Participants | 6 | 6

2. Secondary Outcome: Overall Detection Rate of Prostate Cancer Between Arm A mpMRI+ and Arm B
Description: Number of overall positive prostate cancer (Combined positive and clinically significant positive results) Not all positive prostate biopsies are considered clinically significant. Clinically significant results indicate further work up and/or treatment. Physicians and patients may choose not to just monitor non-clinically significant prostate results for future changes. The overall detection rate will report the total number of both non-clinically significant positive results and clinically significant results.
Time Frame: Within 2-4 wks from biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | MRI/Ultrasound Transperineal Prostate Biopsy | Transrectal Ultrasound-guided Prostate Biopsy
Number analyzed (Participants) | 9 | 11
Participants | 8 | 7

3. Secondary Outcome: Comparison of UTI Incidence in Arm A mpMRI+ and Arm B
Description: Number of confirmed UTIs
Time Frame: From the time of biopsy through 4 weeks post-biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | MRI/Ultrasound Transperineal Prostate Biopsy | Transrectal Ultrasound-guided Prostate Biopsy
Number analyzed (Participants) | 9 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Time of biopsy through 2 to 4 weeks post biopsy
Arm/Group | MRI/Ultrasound Transperineal Prostate Biopsy | Transrectal Ultrasound-guided Prostate Biopsy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03044197/Prot_SAP_000.pdf